CLINICAL TRIAL: NCT02589782
Title: A Randomised, Controlled, Open-Label, Phase II-III Trial to Evaluate the Safety and Efficacy of Regimens Containing Bedaquiline and Pretomanid for the Treatment of Adult Patients With Pulmonary Multidrug Resistant Tuberculosis
Brief Title: Pragmatic Clinical Trial for a More Effective Concise and Less Toxic MDR-TB Treatment Regimen(s)
Acronym: TB-PRACTECAL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medecins Sans Frontieres, Netherlands (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Global Alliance for TB Drug Development (Other); University College, London (Other); Drugs for Neglected Diseases (Other); Swiss Tropical & Public Health Institute (Other); eResearch Technology, Inc. (Industry); Ministry of Health, Republic of Uzbekistan (Other Government); World Health Organization (Other); Ministry of Public Health, Republic of Belarus (Other Government); THINK TB & HIV Investigative Network (Network); University of Liverpool (Other); Wits Health Consortium (Pty) Ltd (Other); Rutgers, The State University of New Jersey (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1541
Record Dates: First submitted 2015-10-15; First posted 2015-10-28 (Estimated); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Tuberculosis, Multidrug-Resistant; Extensively Drug-Resistant Tuberculosis; Tuberculosis, Pulmonary
Keywords: bedaquiline; Nitroimidazoles; diarylquinolines; linezolid; clofazimine; pretomanid; moxifloxacin
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Extensively Drug-Resistant Tuberculosis; Tuberculosis, Pulmonary | interventions — bedaquiline; pretomanid; Moxifloxacin; Linezolid; Clofazimine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Regimen 1 (Experimental): Bedaquiline: 400 mg once daily for 2 weeks followed by 200 mg 3 times per week for 22 weeks Pretomanid: 200mg once daily for 24 weeks Moxifloxacin: 400 mg once daily for 24 weeks Linezolid: 600mg daily for 16 weeks then 300mg daily (or 600mg x3/wk) for the remaining 8 weeks or earlier when moderately tolerated
  Interventions: Drug: Bedaquiline; Drug: Pretomanid; Drug: Moxifloxacin; Drug: Linezolid
- Regimen 2 (Experimental): Bedaquiline: 400 mg once daily for 2 weeks followed by 200 mg 3 times per week for 22 weeks Pretomanid: 200mg once daily for 24 weeks Linezolid: 600mg daily for 16 weeks then 300mg daily (or 600mg x3/wk) for the remaining 8 weeks or earlier when moderately tolerated Clofazimine: 50 mg (less than 33 kg), 100 mg (more than 33 kg) for 24 weeks
  Interventions: Drug: Bedaquiline; Drug: Pretomanid; Drug: Linezolid; Drug: Clofazimine
- Regimen 3 (Experimental): Bedaquiline: 400 mg once daily for 2 weeks followed by 200 mg 3 times per week for 22 weeks Pretomanid: 200mg once daily for 24 weeks Linezolid: 600mg daily for 16 weeks then 300mg daily (or 600mg x3/wk) for the remaining 8 weeks or earlier when moderately tolerated)
  Interventions: Drug: Bedaquiline; Drug: Pretomanid; Drug: Linezolid
- Control Regimen (Active Comparator): Locally accepted standard of care which is consistent with the WHO recommendations for the treatment of M/XDR-TB.
  Interventions: Drug: Locally accepted standard of care which is consistent with the WHO recommendations for the treatment of M/XDR-TB.

INTERVENTIONS:
Drug: Bedaquiline
  Other Names: Sirturo; R207910; TMC207
  Arms: Regimen 1; Regimen 2; Regimen 3
Drug: Pretomanid
  Other Names: PA-824
  Arms: Regimen 1; Regimen 2; Regimen 3
Drug: Moxifloxacin
  Other Names: Avelox
  Arms: Regimen 1
Drug: Linezolid
  Other Names: Zyvox
  Arms: Regimen 1; Regimen 2; Regimen 3
Drug: Clofazimine
  Other Names: Lamprene
  Arms: Regimen 2
Drug: Locally accepted standard of care which is consistent with the WHO recommendations for the treatment of M/XDR-TB.
  Arms: Control Regimen

SUMMARY:
TB PRACTECAL is a multi-centre, open label, multi-arm, randomised, controlled, phase II-III trial; evaluating short treatment regimens containing bedaquiline and pretomanid in combination with existing and re-purposed anti-TB drugs for the treatment of biologically confirmed pulmonary multi drug-resistant TB (MDR-TB).

DETAILED DESCRIPTION:
This is a multi-centre, open label, multi-arm, randomised, controlled, phase II-III trial; evaluating short treatment regimens containing bedaquiline and pretomanid in combination with existing and re-purposed anti-TB drugs for the treatment of biologically confirmed pulmonary multidrug-resistant TB (MDR-TB).

The study will be divided into two stages, with a seamless transition between the stages, meaning recruitment into an arm will only stop after a decision has been taken following stage 1 primary end point data analysis. All recruited patients will be followed up to 108 weeks post randomisation unless they die or withdraw consent. The local standard of care (SOC) MDR-TB regimen will be used as the internal control for both safety and efficacy.

The first stage corresponds to a Phase II trial of safety and preliminary efficacy in patients with MDR-TB. Patients will be recruited into 3 parallel B and Pa containing regimen arms plus a SOC control. The main objective of Stage 1 is to select drug regimens for evaluation in Stage 2 based on 8 week safety and efficacy endpoints. All stage 1 patients will be hospitalised for 8 weeks for intensive cardiological evaluations to establish the QT-specific liability of the regimens.

Investigational arms that do not meet predefined safety and efficacy criteria (percentage culture conversion >40%; percentage discontinuation and death <45%) will not be considered for further evaluation. The regimens that do not meet these pre-defined safety and/or efficacy criteria will be eligible to be evaluated for long term safety, tolerability and efficacy in Stage 2.

If less than two investigational arms are available for stage two assessment, the SAC will make recommendations on whether new arms should be introduced in the study. If more than two arms are available for the Stage 2 assessment, two regimens will be chosen. The SAC will make recommendations on which arms to take forward to the trial steering committee.

The second stage corresponds to a phase III trial. Patients in this stage will be recruited into the arms chosen from stage 1 plus the SOC. The regimens will primarily be evaluated for safety and efficacy in comparison with the SOC arm at 72 weeks post randomisation. The primary efficacy outcome will be a composite endpoint of the percentage of unfavourable outcomes. The secondary outcomes will include safety outcomes and in particular the percentage of Grade 3 or 4 AEs and SAEs in the investigational regimens compared with the SOC.

ELIGIBILITY:
Inclusion criteria:

Patients eligible for inclusion in the trial must fulfil all of the following criteria:

* Male or female subjects aged 15 years of age or above, regardless of HIV status;
* Microbiological test (molecular or phenotypic) confirming presence of M. tuberculosis;
* Resistant to at least rifampicin by either molecular or phenotypic drug susceptibility test;
* Completed informed consent form (ICF);

Exclusion criteria:

Patients will not be eligible for inclusion in the trial if they meet any of the following criteria:

* Known allergies, hypersensitivity, or intolerance to any of the study drugs;
* Pregnant or breast-feeding; or unwilling to use appropriate contraceptive measures
* Liver enzymes >3 times the upper limit of normal (AST or ALT);
* Any condition (social or medical) which, in the opinion of the investigator, would make study participation unsafe;
* Taking any medications contraindicated with the medicines in the trial;
* QTcF > 450ms;
* One or more risk factors for QT prolongation (excluding age and gender) or other uncorrected risk factors for TdP;
* History of cardiac disease, syncopal episodes, symptomatic or asymptomatic arrhythmias (with the exception of sinus arrhythmia);
* Any baseline biochemical laboratory value consistent with Grade 4 toxicity.
* Moribund
* Known resistance to bedaquiline, pretomanid, delamanid or linezolid.
* Prior use of bedaquiline and/or pretomanid and/or linezolid and/or delamanid for one or more months.
* Patients not eligible to start a new course of MDR-TB/XDR-TB treatment according to local protocol, including but not limited to:

  * currently on MDR-TB treatment for more than 2 weeks (and not failing)
  * unstable address
  * loss to follow-up in previous treatment with no change in circumstance and motivation.
* Tuberculous meningoencephalitis, brain abscesses, osteomyelitis or arthritis.

PKPD inclusion/exclusion:

* Adult patients (aged 18 years or above) recruited into the investigational arms of the TB-PRACTECAL trial in the approved sites.
* Willing to sign the sub-study informed consent form after agreeing to the additional blood draws.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Stage 1:Percentage of patients with culture conversion in liquid media at 8 weeks post randomisation. | 8 weeks post randomisation
Stage 1: Percentage of patients who discontinue treatment for any reason or die | 8 weeks post randomisation
Stage 2: Percentage of patients with an unfavourable outcome (failure, death, recurrence, loss to follow-up) | 72 weeks post-randomisation

SECONDARY OUTCOMES:
Stage 1: Percentage of patients with grade 3 or higher QT prolongation | within 8 weeks post randomisation
Stage 1: Percentage of patients experiencing at least one Serious Adverse Event (SAE) | within 8 weeks post randomisation
Stage 1:Percentage of patients experiencing at least one new grade 3 or higher Adverse Event | within 8 weeks post randomisation
Stage 2: Percentage of patients with culture conversion | 12 weeks post randomisation
Stage 2: Percentage of patients with an unfavourable outcome (i.e. failure, treatment discontinuation, death, loss to follow up) | 24 weeks post randomisation
Stage 2: Percentage of patients with an unfavourable outcome (i.e. failure, treatment discontinuation, death, loss to follow up, still on treatment at censure and recurrence) | 108 weeks post randomisation
Stage 2: Median time to culture conversion | 108 weeks
Stage 2: Percentage of patients with an SAE or new grade 3 or higher AE | 72 weeks post randomisation
Stage 2: Percentage of patients with an SAE or new grade 3 or higher AE | 108 weeks post randomisation
Stage 2: Percentage of patients with an SAE or new grade 3 or higher AE at the end of treatment | 24 weeks in investigational arms and 108 weeks in SOC arm
  The percentage of patients with an SAE or new grade 3 or higher AE at the end of treatment in the investigational arms (maximum of 24 weeks) and the SOC arm which varies in length (maximum 108 weeks).
Stage 2: Mean single ΔQTcF | 24 weeks post randomisation
Stage 2: Percentage of patients experiencing recurrence | week 48 in investigational arms
Stage 2: Plasma drug concentrations | In relation to dose intake and start of treatment over a 72 week period
Stage 2: TB drug hair levels | In relation to dose intake and start of treatment over a 72 week period

CONTACTS AND LOCATIONS:
Overall Officials: Bern-Thomas Nyang'wa, MD, Principal Investigator — Medecins Sans Frontieres, Netherlands
Locations (7):
- Republican Scientific and Practical Centre for Pulmonology and Tuberculosis hospital, Minsk, Belarus
- South Africa (4):
  - Helen Jospeh Hospital, Johannesburg, Gauteng
  - THINK Clinical Trial Unit, Hillcrest, Durban, KwaZulu-Natal
  - King DinuZulu Hospital, Durban, KwaZulu-Natal
  - Doris Goodwin Hospital, Pietermaritzburg, KwaZulu-Natal
- Uzbekistan (2):
  - Republican TB Hospital No. 2, Nukus, Karakalpakstan
  - Sh Alimov Republican Specialised Scientific-Practical Medical Centre for Phthysiology and Pulmonology Hospital, Tashkent

IPD SHARING:
Plan to Share IPD: Yes
Deidentified dataset will be made available via the TB-PACTS repository.
Supporting Information: Study Protocol, SAP
Time Frame: Q3 2024
URL: https://c-path.org/tools-platforms/tb-pacts/

REFERENCES:
- [Derived] Motta I, Cusinato M, Ludman AJ, Lachenal N, Dodd M, Soe M, Abdrasuliev T, Usmanova R, Butabekov I, Nikolaevna TZ, Liverko I, Parpieva N, Moodliar R, Solodovnikova V, Kazounis E, Nyang'wa B-T, Fielding KL, Berry C. How much should we still worry about QTc prolongation in rifampicin-resistant tuberculosis? ECG findings from TB-PRACTECAL clinical trial. Antimicrob Agents Chemother. 2024 Jul 9;68(7):e0053624. doi: 10.1128/aac.00536-24. Epub 2024 Jun 6. PMID 38842323
- [Derived] Nyang'wa BT, Berry C, Kazounis E, Motta I, Parpieva N, Tigay Z, Moodliar R, Dodd M, Solodovnikova V, Liverko I, Rajaram S, Rassool M, McHugh T, Spigelman M, Moore DA, Ritmeijer K, du Cros P, Fielding K; TB-PRACTECAL team. Short oral regimens for pulmonary rifampicin-resistant tuberculosis (TB-PRACTECAL): an open-label, randomised, controlled, phase 2B-3, multi-arm, multicentre, non-inferiority trial. Lancet Respir Med. 2024 Feb;12(2):117-128. doi: 10.1016/S2213-2600(23)00389-2. Epub 2023 Nov 16. PMID 37980911
- [Derived] Nyang'wa BT, Berry C, Kazounis E, Motta I, Parpieva N, Tigay Z, Solodovnikova V, Liverko I, Moodliar R, Dodd M, Ngubane N, Rassool M, McHugh TD, Spigelman M, Moore DAJ, Ritmeijer K, du Cros P, Fielding K; TB-PRACTECAL Study Collaborators. A 24-Week, All-Oral Regimen for Rifampin-Resistant Tuberculosis. N Engl J Med. 2022 Dec 22;387(25):2331-2343. doi: 10.1056/NEJMoa2117166. PMID 36546625
- [Derived] Berry C, du Cros P, Fielding K, Gajewski S, Kazounis E, McHugh TD, Merle C, Motta I, Moore DAJ, Nyang'wa BT. TB-PRACTECAL: study protocol for a randomised, controlled, open-label, phase II-III trial to evaluate the safety and efficacy of regimens containing bedaquiline and pretomanid for the treatment of adult patients with pulmonary multidrug-resistant tuberculosis. Trials. 2022 Jun 13;23(1):484. doi: 10.1186/s13063-022-06331-8. PMID 35698158